CLINICAL TRIAL: NCT04123405
Title: Efficacy and Safety of Acetylcysteine for the Treatment of Acute Uncomplicated Rhinosinusitis: a Prospective, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Acetylcysteine for the Treatment of Acute Uncomplicated Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-08-EFT-1; 2019-000060-20 (EudraCT Number)
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Rhinosinusitis
Keywords: acute uncomplicated rhinosinusitis, acetylcysteine
MeSH Terms: conditions — Rhinosinusitis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: 600 mg acetylcysteine (Experimental): one tablet test product plus three tablets placebo per day (taken as two tablets dissolved in a glass of water, twice daily)
  Interventions: Drug: acetylcysteine; Drug: Placebo
- Group B: 1200 mg acetylcysteine (Experimental): two tablets test product plus two tablets placebo per day (taken as two tablets dissolved in a glass of water, twice daily)
  Interventions: Drug: acetylcysteine; Drug: Placebo
- Group C: 2400 mg acetylcysteine (Experimental): four tablets test product per day (taken as two tablets dissolved in a glass of water, twice daily)
  Interventions: Drug: acetylcysteine
- Group D: Placebo (Placebo Comparator): four tablets placebo per day (taken as two tablets dissolved in a glass of water, twice daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: acetylcysteine — 600 mg tablet
  Arms: Group A: 600 mg acetylcysteine; Group B: 1200 mg acetylcysteine; Group C: 2400 mg acetylcysteine
Drug: Placebo — Placebo to acetylcysteine
  Arms: Group A: 600 mg acetylcysteine; Group B: 1200 mg acetylcysteine; Group D: Placebo

SUMMARY:
The trial was conducted as a prospective, randomized, multinational, multicenter, double-blind study in 4 parallel groups of patients.

DETAILED DESCRIPTION:
The study was the prospective, randomized, multinational, multicenter, double-blind study in 4 parallel groups of patients.

Patients underwent screening examinations at Visit 1. Patients who met all inclusion/ no exclusion criteria were randomized at the baseline visit (Day 1) to the double-blind treatment for a duration of 14 days but in case of delayed final visit (Day 15) the patient could voluntarily take reserve study medication for a maximum of 3 additional days.

After the end of the double-blind treatment phase, the patients underwent an end-of-treatment (EOT) examinations on Day 15 (+3).

A follow-up phone call within 7 days after Day 15 (or earlier in case of premature termination) was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 14 and 75 years inclusive on the date of consent
2. Diagnosis of acute, uncomplicated rhinosinusitis defined at screening visit 1 and at Visit 2 as:

   1. major symptom score (MSS) assessed by the patient ≥8 and ≤12 points for the following: rhinorrhea/ anterior discharge, postnasal drip, nasal congestion, headache, and facial pain/pressure, whereupon the nasal congestion is mandatory and no more than 3 of the 5 symptoms are rated as severe
   2. individual score for facial pain/pressure ≥1 (mild) and ≤2 (moderate)
   3. presence of symptoms ≤3 days prior to screening visit
3. For adults (≥18 years): Informed consent to participate in the trial provided in written form; For adolescents (≥14 - <18 years): own subject informed consent/ assent to participate in the trial and the informed consent from all parent(s)/ legal guardian(s) provided in written form.

Exclusion Criteria:

1. History of hypersensitivity or intolerance to the active substance or any of the excipients of the trial medication
2. Patient with history of hereditary fructose intolerance, galactose intolerance, lactase deficiency or glucose-galactose malabsorption
3. Chronic rhinosinusitis (symptoms lasting longer than 3 months)
4. Subjects who have undergone sinus or nasal surgery for chronic rhinosinusitis in the 6 months prior to screening visit
5. Sinus lavage within 7 days prior to screening visit
6. Odontogenic rhinosinusitis
7. Allergic (perennial or seasonal) rhinitis
8. Bronchial asthma or chronic obstructive pulmonary disease
9. Nasal polyposis or clinically relevant nasal septum deviation
10. Concomitant otitis
11. Intranasal or systemic use of corticosteroids within 30 days prior to screening visit
12. Intranasal or systemic use of antibiotics within 30 days prior to screening visit
13. Use of nasal decongestants within 2 days prior to screening visit
14. Concomitant treatment of common cold-like symptoms within 7 days prior to screening visit with any of the following:

    1. Analgesics
    2. Non-steroidal anti-inflammatory drugs
    3. Antihistamines
15. Concomitant use of intranasal saline irrigation
16. Use of immunosuppressive agents within 30 days prior to screening visit
17. Immunocompromised state
18. Suspicion for acute bacterial rhinosinusitis (defined as presence of purulence for 3 to 4 days with fever ≥ 38.3°C)
19. Pregnant or breast-feeding female patient
20. Female patient of childbearing potential (not surgically sterilized/hysterectomized or postmenopausal for at least 1 year) who is not currently using (documented at screening visit) and not willing to use medically reliable methods of contraception for the entire trial duration such as oral, injectable or implantable contraceptives, intrauterine contraceptive devices (IUD), sexual abstinence or vasectomized partner
21. Any other condition of the patient (e.g. serious or unstable medical or psychological condition, acute psychosis) that in the opinion of the investigator may compromise evaluation of the trial treatment or may jeopardize patient's safety, compliance or adherence to protocol requirements
22. Participation in ANY research study involving another investigational medicinal product (IMP) within 30 days prior to screening visit, or simultaneous participation in another clinical study or previous participation in present study
23. Suspected alcohol/ drug dependence or abuse (including heavy smoking: ≥ 20 cigarettes daily)
24. Use of snuff tobacco
25. Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of the trial
26. Subjects who are known or suspected:

    * not to comply with the trial directives
    * not to be reliable or trustworthy
    * to be a dependent person, e.g. a relative, family member, or member/employee of the investigator's or sponsor's staff
    * subject is in custody or submitted to an institution due to a judicial order.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 944 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (19):
- Bulgaria (6):
  - Sandoz Investigative Site, Burgas
  - Sandoz Investigative Site, Gabrovo
  - Sandoz Investigative Site, Plovdiv
  - Sandoz Investigative Site, Sliven
  - Sandoz Investigative Site, Sofia
  - Sandoz Investigative Site, Yambol
- Germany (3):
  - Sandoz Investigative Site, Aachen
  - Sandoz Investigative Site, Dresden
  - Sandoz Investigative Site, Duisburg
- Moldova (2):
  - Sandoz Investigative Site, Chisinau
  - Sandoz Investigative Site, Orhei
- Russia (8):
  - Sandoz Investigative Site, Kazan'
  - Sandoz Investigative Site, Kemerovo
  - Sandoz Investigative Site, Moscow
  - Sandoz Investigative Site, Novosibirsk
  - Sandoz Investigative Site, Ryazan
  - Sandoz Investigative Site, Saint Petersburg
  - Sandoz Investigative Site, Smolensk
  - Sandoz Investigative Site, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 42 clinical centers located in Bulgaria, Germany, Moldova and Russia.
Pre-assignment Details: Participants were randomized in 1:1:1:1 ratio
Period: Overall Study
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Started (Randomized) | 235 | 238 | 238 | 233
Full Analysis Set (all randomized patients who received at least one dose of the trial medication and who had at least one post-baseline assessment of MSS during the double-blind treatment period) | 235 | 236 | 238 | 230
Per-protocol Set (all FAS-evaluable patients who completed the double-blind treatment period without major protocol violations that could affect the efficacy evaluation) | 213 | 215 | 212 | 207
Safety Set (all randomized patients who received at least one dose of the trial medication) | 235 | 238 | 238 | 233
Completed | 231 | 231 | 235 | 225
Not Completed | 4 | 7 | 3 | 8
Not completed — Adverse Event | 1 | 2 | 3 | 3
Not completed — Exclusion criteria met | 1 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 2
Not completed — Contact to subject lost | 0 | 0 | 0 | 1
Not completed — screening failure | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo | Total
Number analyzed (Participants) | 235 | 238 | 238 | 233 | 944
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (13.8) | 40.7 (13.6) | 41.3 (13.1) | 41.1 (14.0) | 41.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 142 | 145 | 141 | 556
  Male | 107 | 96 | 93 | 92 | 388
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 230 | 235 | 232 | 231 | 928
  Asian | 4 | 2 | 5 | 2 | 13
  Unknown | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Daily Major Symptom Score (MSS) Over the Entire Treatment Period, Full Analysis Set
Description: The MSS combines the 5 most relevant symptoms of rhinosinusitis based on expert clinician recommendations (rhinorrhea/ anterior discharge, postnasal drip, nasal congestion, headache, and facial pain/pressure). The patient rated the severity of each of the five symptoms of the MSS using a four-point rating scale of increasing severity (0 = none/not present, 1 = mild, 2 = moderate, 3 = severe). The MSS is then the sum of single ratings with a possible range from 0 to 15.
  Mean change from baseline in the daily Major Symptom Score (MSS) over the entire treatment period was calculated as the average total score from Day 2 to 15 compared to Baseline (Day 1). Negative change from baseline means improvement.
Time Frame: Baseline (Day 1), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: Full-Analysis Set (FAS) included all randomized patients who received at least one dose of the trial medication and who had at least one post-baseline assessment of MSS during the double-blind treatment period.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 235 | 236 | 238 | 230
Score on a scale | -4.8213 (1.98247) | -4.7394 (1.99090) | -4.7758 (1.96938) | -5.0180 (1.98262)

2. Primary Outcome: Mean Change From Baseline in the Daily Major Symptom Score (MSS) Over the Entire Treatment Period, Per-Protocol Set
Description: as for outcome 1
Time Frame: Baseline (Day 1), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: Per-Protocol Set (PPS) included all FAS-evaluable patients who completed the double-blind treatment period without major protocol violations that could affect the efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 213 | 215 | 212 | 207
Score on a scale | -4.9085 (1.92431) | -4.8688 (1.84448) | -4.8002 (1.90569) | -5.1256 (1.95072)

3. Secondary Outcome: Time to Onset of Action, Full Analysis Set
Description: Time to onset of action was defined as first day of active treatment on which MSS showed statistically significant (p value<0.05) improvement from placebo.
Time Frame: Baseline (Day 1), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: as for outcome 1
Measure: Number; unit: Days
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine
Number analyzed (Participants) | 235 | 236 | 238
Days | NA — There was no statistically significant improvement of the drug from placebo on any day | NA — There was no statistically significant improvement of the drug from placebo on any day | NA — There was no statistically significant improvement of the drug from placebo on any day

4. Secondary Outcome: Time to Onset of Action, Per-Protocol Set
Description: as for outcome 3
Time Frame: Baseline (Day 1), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: as for outcome 2
Measure: Number; unit: Days
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine
Number analyzed (Participants) | 213 | 215 | 212
Days | NA — There was no statistically significant improvement of the drug from placebo on any day | NA — There was no statistically significant improvement of the drug from placebo on any day | NA — There was no statistically significant improvement of the drug from placebo on any day

5. Secondary Outcome: Major Symptom Score (MSS) Development Over the Course of the Study, Full Analysis Set
Description: as for outcome 1
Time Frame: Baseline (Day 1), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 235 | 236 | 238 | 230
Score on a scale
  Day 1 (Baseline) | 9.634 (1.1181) | 9.640 (1.0647) | 9.702 (1.0101) | 9.683 (1.0652)
  Day 2 | 9.021 (2.0348) | 9.004 (1.9883) | 9.038 (2.1235) | 9.074 (1.9866)
  Day 3 | 8.485 (2.3376) | 8.513 (2.2303) | 8.416 (2.4390) | 8.609 (2.1298)
  Day 4 | 7.821 (2.4482) | 7.695 (2.5130) | 7.723 (2.7156) | 7.761 (2.5058)
  Day 5 | 6.983 (2.7284) | 6.979 (2.5706) | 7.013 (2.7490) | 6.917 (2.6312)
  Day 6 | 6.323 (2.7807) | 6.203 (2.8719) | 6.315 (2.7980) | 6.039 (2.7838)
  Day 7 | 5.528 (2.9747) | 5.538 (2.7449) | 5.576 (2.8508) | 5.126 (2.7096)
  Day 8 | 4.766 (2.8631) | 4.750 (2.6755) | 4.891 (2.7598) | 4.387 (2.6004)
  Day 9 | 4.204 (2.8149) | 4.322 (2.7254) | 4.445 (2.7381) | 3.839 (2.5924)
  Day 10 | 3.634 (2.6815) | 3.763 (2.6391) | 3.845 (2.6634) | 3.404 (2.6805)
  Day 11 | 3.051 (2.5229) | 3.284 (2.6658) | 3.256 (2.5716) | 2.843 (2.6469)
  Day 12 | 2.609 (2.5200) | 2.754 (2.5680) | 2.756 (2.3795) | 2.413 (2.5608)
  Day 13 | 2.038 (2.4202) | 2.246 (2.5296) | 2.218 (2.4293) | 1.943 (2.4174)
  Day 14 | 1.583 (2.3289) | 1.941 (2.5375) | 1.836 (2.3300) | 1.596 (2.3637)
  Day 15 | 1.332 (2.1485) | 1.614 (2.4459) | 1.634 (2.3178) | 1.352 (2.1882)

6. Secondary Outcome: Major Symptom Score (MSS) Development Over the Course of the Study, Per-protocol Set
Description: as for outcome 1
Time Frame: Baseline (Day 1), Day 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 213 | 215 | 212 | 207
Score on a scale
  Day 1 (Baseline) | 9.657 (1.1201) | 9.628 (1.0595) | 9.698 (1.0319) | 9.676 (1.0823)
  Day 2 | 9.080 (2.0160) | 8.935 (2.0268) | 9.127 (2.0089) | 9.068 (2.0278)
  Day 3 | 8.545 (2.2890) | 8.395 (2.2583) | 8.528 (2.2591) | 8.594 (2.1921)
  Day 4 | 7.803 (2.4779) | 7.577 (2.5472) | 7.816 (2.5849) | 7.739 (2.5750)
  Day 5 | 6.962 (2.7401) | 6.874 (2.5865) | 7.061 (2.6522) | 6.821 (2.6717)
  Day 6 | 6.315 (2.7914) | 6.093 (2.8809) | 6.349 (2.7000) | 5.937 (2.8354)
  Day 7 | 5.479 (2.9550) | 5.400 (2.7151) | 5.604 (2.7800) | 4.981 (2.7163)
  Day 8 | 4.685 (2.8250) | 4.605 (2.6399) | 4.892 (2.7421) | 4.237 (2.5914)
  Day 9 | 4.117 (2.7558) | 4.181 (2.6773) | 4.382 (2.6734) | 3.652 (2.5495)
  Day 10 | 3.521 (2.6127) | 3.628 (2.5174) | 3.741 (2.5507) | 3.222 (2.6197)
  Day 11 | 2.934 (2.4039) | 3.144 (2.5214) | 3.146 (2.4538) | 2.705 (2.6042)
  Day 12 | 2.493 (2.3485) | 2.572 (2.3785) | 2.608 (2.2228) | 2.300 (2.4902)
  Day 13 | 1.897 (2.2146) | 2.065 (2.2949) | 2.085 (2.2013) | 1.816 (2.3077)
  Day 14 | 1.432 (2.0812) | 1.749 (2.2779) | 1.708 (2.1128) | 1.444 (2.2198)
  Day 15 | 1.221 (1.9530) | 1.409 (2.1312) | 1.524 (2.0846) | 1.193 (1.9636)

7. Secondary Outcome: Sino-Nasal Outcome Test (SNOT-22) by Visit, Full Analysis Set
Description: SNOT-22 Questionnaire is a disease specific Health-Related Quality of Life (HRQoL) measure that comprises a list of 22 symptoms and social or emotional consequences of the nasal disorder. Every participant is asked to rate how severe each problem had been on a scale from 0 (no problem) to 5 (problem as bad as it can be). The total score is the sum of the scores for all 22 items, ranging from 0 to 110, with a lower score indicating better HRQoL.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 235 | 236 | 238 | 230
Score on a scale
  Day 1 (Baseline): number analyzed (Participants) | 209 | 213 | 212 | 203
  Day 1 (Baseline) | 37.8 (16.89) | 36.3 (15.82) | 36.7 (16.21) | 36.3 (17.00)
  Day 7: number analyzed (Participants) | 210 | 211 | 215 | 205
  Day 7 | 23.6 (15.01) | 21.2 (13.14) | 22.3 (13.95) | 21.1 (13.56)
  Day 14: number analyzed (Participants) | 210 | 211 | 216 | 208
  Day 14 | 7.2 (10.80) | 6.9 (11.15) | 7.0 (10.07) | 6.5 (10.28)

8. Secondary Outcome: Sino-Nasal Outcome Test (SNOT-22) by Visit, Per Protocol Set
Description: as for outcome 7
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 213 | 215 | 212 | 207
Score on a scale
  Day 1 (Baseline): number analyzed (Participants) | 193 | 197 | 194 | 188
  Day 1 (Baseline) | 37.7 (16.64) | 36.7 (15.89) | 36.4 (15.86) | 36.2 (16.88)
  Day 7: number analyzed (Participants) | 195 | 196 | 194 | 190
  Day 7 | 23.3 (14.92) | 21.2 (13.32) | 22.2 (14.27) | 21.0 (13.78)
  Day 14: number analyzed (Participants) | 195 | 198 | 194 | 193
  Day 14 | 6.9 (10.49) | 7.1 (11.43) | 6.8 (9.67) | 6.6 (10.50)

9. Secondary Outcome: Sino-Nasal Outcome Test (SNOT-22) by Change to Baseline, Full Analysis Set
Description: SNOT-22 Questionnaire is a disease specific Health-Related Quality of Life (HRQoL) measure that comprises a list of 22 symptoms and social or emotional consequences of the nasal disorder. Every participant is asked to rate how severe each problem had been on a scale from 0 (no problem) to 5 (problem as bad as it can be). The total score is the sum of the scores for all 22 items, ranging from 0 to 110, with a lower score indicating better HRQoL. A negative change from baseline in SNOT-22 is considered a favorable outcome.
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 235 | 236 | 238 | 230
Score on a scale
  Day 7: number analyzed (Participants) | 207 | 210 | 211 | 201
  Day 7 | -35.8 (33.25) | -38.2 (37.48) | -36.7 (34.61) | -39.6 (30.42)
  Day 14: number analyzed (Participants) | 204 | 209 | 209 | 201
  Day 14 | -79.3 (31.27) | -78.9 (31.11) | -78.6 (30.53) | -81.5 (26.54)

10. Secondary Outcome: Sino-Nasal Outcome Test (SNOT-22) by Change to Baseline, Per Protocol Set
Description: as for outcome 9
Time Frame: Baseline (Day 1), Day 7 and Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 213 | 215 | 212 | 207
Score on a scale
  Day 7: number analyzed (Participants) | 192 | 195 | 193 | 188
  Day 7 | -36.4 (32.64) | -39.5 (36.68) | -36.7 (33.44) | -39.6 (30.60)
  Day 14: number analyzed (Participants) | 189 | 196 | 192 | 188
  Day 14 | -79.8 (30.90) | -78.6 (31.77) | -79.1 (30.16) | -81.0 (27.10)

11. Secondary Outcome: Number of Responders and Non-responders to Treatment, Full Analysis Set
Description: Number of responders and non-responders to treatment based on the assessment of overall response to treatment by the investigator were reported.
Time Frame: Day 4, 7, 10 and 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 235 | 236 | 238 | 230
Participants
  Day 4: number analyzed (Participants) | 233 | 235 | 237 | 229
  Day 4: Responders | 148 | 152 | 151 | 150
  Day 4: Non-responders | 85 | 83 | 86 | 79
  Day 7: number analyzed (Participants) | 232 | 235 | 227 | 227
  Day 7: Responders | 209 | 206 | 212 | 209
  Day 7: Non-responders | 23 | 29 | 15 | 18
  Day 10: number analyzed (Participants) | 231 | 232 | 235 | 225
  Day 10: Responders | 225 | 225 | 230 | 219
  Day 10: Non-responders | 6 | 7 | 5 | 6
  Day 15: number analyzed (Participants) | 234 | 232 | 238 | 228
  Day 15: Responders | 230 | 226 | 230 | 224
  Day 15: Non-responders | 4 | 6 | 8 | 4

12. Secondary Outcome: Number of Responders and Non-responders to Treatment, Per-Protocol Set
Description: as for outcome 11
Time Frame: Day 4, 7, 10 and 15
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
Number analyzed (Participants) | 213 | 215 | 212 | 207
Participants
  Day 4: Responders | 138 | 140 | 132 | 134
  Day 4: Non-responders | 75 | 75 | 80 | 73
  Day 7: Responders | 192 | 190 | 191 | 192
  Day 7: Non-responders | 21 | 25 | 21 | 15
  Day 10: Responders | 207 | 210 | 209 | 202
  Day 10: Non-responders | 6 | 5 | 3 | 5
  Day 15: Responders | 211 | 210 | 206 | 205
  Day 15: Non-responders | 2 | 5 | 6 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment up to maximum duration of 22 days.
Description: Any signs or symptoms were collected from first dose of study treatment up to maximum duration of 22 days.
Arm/Group | Group A: 600 mg Acetylcysteine | Group B: 1200 mg Acetylcysteine | Group C: 2400 mg Acetylcysteine | Group D: Placebo
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/238 | 0/238 | 0/233
Serious Adverse Events (participants affected / at risk) | 0/235 | 0/238 | 0/238 | 1/233
Other Adverse Events (participants affected / at risk) | 9/235 | 15/238 | 15/238 | 8/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: 600 mg Acetylcysteine (N=235) | Group B: 1200 mg Acetylcysteine (N=238) | Group C: 2400 mg Acetylcysteine (N=238) | Group D: Placebo (N=233)
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: 600 mg Acetylcysteine (N=235) | Group B: 1200 mg Acetylcysteine (N=238) | Group C: 2400 mg Acetylcysteine (N=238) | Group D: Placebo (N=233)
Ear congestion (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 1 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1
Human chorionic gonadotropin increased (Investigations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT04123405/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT04123405/SAP_001.pdf